CLINICAL TRIAL: NCT03277235
Title: Effectiveness of a Resilience Model-Based Cancer Prehabilitation Program for Patients With Newly Diagnosed Colorectal Cancer: A Randomized Controlled Trial
Brief Title: Effect of a Resilience Model-Based Program for Patients With Newly Diagnosed Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201612224RIND
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Cancer (MSI-H)
Keywords: resilience; cancer prehabilitation; physical distress; psychological distress; spiritual well-being; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resilience model-based cancer prehabilitation program plus standard care (Experimental): 12-week care plan with 5 in-person and 12 remote sessions, including both physical and psychological components.
  Interventions: Behavioral: Resilience model-based total care plan
- Control (Other): standard care
  Interventions: Behavioral: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Resilience model-based total care plan — 12-week care plan with 5 times face-to-face intervention and weekly phone call follow-up to increase the protective factors (positive thinking. problem-solving, finding meaning, and social connection) and decrease the risk factors (disease-related distress and defense coping) of resilience
  Arms: Resilience model-based cancer prehabilitation program plus standard care
Behavioral: Standard Care (in control arm) — standard care
  Arms: Control

SUMMARY:
To develop a resilience model-based cancer prehabilitation program and evaluate its efficacy in improving resilience, alleviating symptoms, and enhancing spiritual well-being in patients with newly diagnosed colorectal cancer.

DETAILED DESCRIPTION:
Develop and evaluate the effect of a resilience model-based total care plan on reducing fear of recurrence and GI symptom distress, resilience and improving spiritual well-being in this population.

ELIGIBILITY:
The inclusion criteria were as follows: being aged ≧ 20 years, receiving a new diagnosis of stage 0-III colorectal cancer and being scheduled to undergo surgery, being aware of the diagnosis, being able to communicate in Mandarin or Taiwanese, and providing written informed consent. The exclusion criteria were as follows: receiving a diagnosis of stage IV colorectal cancer, having recurrent colorectal cancer or multiple cancers, and having a history of psychiatric disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Resilience scale | Change from baseline resilience at 12 months
  The questionnaire includes 25 items to assess levels of resilience

SECONDARY OUTCOMES:
Symptom Severity Scale | Change from baseline symptom at 12 months
  The questionnaire includes 24 items to assess symptom severity
Fatigue Symptom Inventory | Change from baseline fatigue at 12 months
  The questionnaire includes 14 items to assess fatigue
Center for Epidemiological Studies Depression Scale | Change from baseline depressive symptoms at 12 months
  The questionnaire includes 20 items to assess depressive symptoms
Fear of Cancer Recurrence Inventory-Short Form | Change from baseline fear of cancer recurrence at 12 months
  The questionnaire includes 9 items to assess fear of cancer recurrence
Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Scale | Change from baseline spiritual well-being at 12 months
  The questionnaire includes 12 items to assess spiritual well-being

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PHD, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chou YJ, Lee YH, Lin BR, Jiang JK, Yang HY, Lin HY, Shun SC. Serial multiple mediation model of fear of cancer recurrence in patients with colorectal cancer. Health Psychol. 2025 Oct;44(10):955-962. doi: 10.1037/hea0001483. Epub 2025 Apr 14. PMID 40232818
- [Derived] Liao YT, Chou YJ, Wu CT, Liu YH, Liang JT, Lai F, Shun SC. Wearable mobile health device for monitoring postoperative ambulation among patients with colorectal cancer undergoing minimally invasive surgery: A prospective comparison study. Int J Med Robot. 2024 Apr;20(2):e2626. doi: 10.1002/rcs.2626. PMID 38517612
- [Derived] Chou YJ, Lin HY, Cooper BA, Lin BR, Jiang JK, Yang HY, Miaskowski C, Shun SC. A Resilience Model for Patients With Colorectal Cancer: A Structural Equation Modeling Analysis. Cancer Nurs. 2022 Jan-Feb 01;45(1):E83-E90. doi: 10.1097/NCC.0000000000000882. PMID 34870940